CLINICAL TRIAL: NCT02176746
Title: Study of Cancer Stem Cell Vaccine That as a Specific Antigen in Metastatic Adenocarcinoma of the Colorectal
Brief Title: A Phase I/II Study of Active Immunotherapy With Cancer Stem Cells Vaccine for Colorectal Cancer
Acronym: CSC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLC-001
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2014-06

CONDITIONS: Neoplasms,Colorectal
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- non-cancer stem cell vaccine (Placebo Comparator): This is no cancer stem cells vaccine in this group
  Interventions: Biological: cancer stem cell vaccine
- giving low dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine
- giving middle dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine
- giving high dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine

INTERVENTIONS:
Biological: cancer stem cell vaccine

SUMMARY:
Most studies of cancer stem cells (CSC) involve the inoculation of cells from human tumors into immunosuppressed mice, preventing an assessment on the immunologic interactions and effects of CSCs. In this study, the investigators examined the vaccination effects produced by CSC-enriched populations from histologically distinct murine tumors after their inoculation into different syngeneic immunocompetent hosts. Enriched CSCs were immunogenic and more effective as an antigen source than unselected tumor cells in inducing protective antitumor immunity.Immune sera from CSC-vaccinated hosts contained high levels of IgG which bound to CSCs, resulting in CSC lysis in the presence of complement.CTLs generated from peripheral blood mononuclear cells or splenocytes harvested from CSC-vaccinated hosts were capable of killing CSCs in vitro. Mechanistic investigations established that CSC-primed antibodies and T cells were capable of selective targeting CSCs and conferring anti-tumor immunity.

DETAILED DESCRIPTION:
To assess the feasibility of generating CSC-loaded DC vaccines for clinical use, the investigators will harvest peripheral blood and tumor specimen from patients with colorectal cancer. The investigators will purify T, B cells and generate DCs from the PBMCs of the colorectal cancer patient.On the other hand, investigators will isolate ALDHhigh and ALDHlow tumor cells from the tumor specimen of the colorectal cancer patient using a similar protocol as investigators reported .

Aim 1: To demonstrate, in vitro, the relative cellular anti-colorectal cancer CSC immunity induced by colorectal cancer CSC-DC primed cytotoxic T cells.

Aim 2: To determine, in vitro, specific binding and lysis of colorectal cancer CSCs by antibodies produced by purified B cells from PBMCs stimulated with colorectal cancer CSC-DC.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 and over
2. Performance status:Karnofsky 70-100%
3. Life expectancy:Greater than 6 months
4. Hematopoietic:Absolute neutrophil count at least 1000/mm 3,Hemoglobin at least 9 g/dL,Platelet count at least 100,000/mm^3
5. Hepatic:Bilirubin less than 2.0 mg/dL No chronic or acute hepatic disease Renal:Creatinine less than 2.5 mg/dL
6. Cardiovascular:

   No chronic or acute cardiac disease (New York Heart Association class III or IV)
7. Pulmonary:

No chronic or acute pulmonary illness such as asthma or chronic obstructive pulmonary disease

Exclusion Criteria:

1. Patients receiving anticoagulation therapy.
2. Patients receiving any other investigational agents.
3. Patients who test positive for Hepatitis B virus, Hepatitis C virus or HIV. 4、level 3 hypertension; 5、severe coronary disease; 6、 myelosuppression; 7、 respiratory disease; 8、 brain metastasis; 9、 chronic infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The number of participants with adverse events | up to 3 months

SECONDARY OUTCOMES:
The secondary objectives are to evaluate vaccine immune responses to the immunizations by the data of body measurements | 1 month

OTHER OUTCOMES:
The dose of CSC vaccine | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Ning N, Pan Q, Zheng F, Teitz-Tennenbaum S, Egenti M, Yet J, Li M, Ginestier C, Wicha MS, Moyer JS, Prince ME, Xu Y, Zhang XL, Huang S, Chang AE, Li Q. Cancer stem cell vaccination confers significant antitumor immunity. Cancer Res. 2012 Apr 1;72(7):1853-64. doi: 10.1158/0008-5472.CAN-11-1400. PMID 22473314
- See also: Related Info — http://www.fudahospital.com/